CLINICAL TRIAL: NCT00001460
Title: Evaluation and Therapy of Heart Disease in Patients Not Participating in Research (Teaching Protocol)
Brief Title: Evaluation and Treatment of Heart Disease in Patients Not Participating in Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950051; 95-H-0051
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2002-04

CONDITIONS: Arrhythmia; Congenital Heart Defect; Heart Disease
Keywords: Training Protocol; Cardiac Diagnosis; Congenital Heart Disease; Acquired Heart Disease; Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Defects, Congenital; Heart Diseases | interventions — Therapeutics

INTERVENTIONS:
Behavioral: inpatient evaluation and management

SUMMARY:
There is an important need to maintain clinical skills, provide quality training and expertise, and provide an environment that stimulates ideas for clinical research.

This study permits inpatient evaluation and management of patients with heart disease who do not qualify to participate in studies currently being conducted by the Cardiology Branch of the National Heart, Lung, and Blood Institute.

DETAILED DESCRIPTION:
There is an important need to maintain clinical skills, to ensure adequate training and expertise, and provide an environment that stimulates ideas for clinical research. This protocol permits inpatient evaluation and management of patients with heart disease who do not fulfill criteria for participation in existing Cardiology Branch research protocols.

ELIGIBILITY:
Patients with signs or symptoms of heart disease.

Patients selected because of either medical or research interest to the Principal Investigator.

Patients must not have unstable angina pectoris, unstable course following recent (within one month) myocardial infarction.

Must not be in New York Heart Association functional class IV heart failure.

A positive pregnancy test will obviate any cardiovascular testing requiring ionizing radiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-01; Study Completion 2002-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States